CLINICAL TRIAL: NCT02748603
Title: Appropriateness of Coronary Angioplasty in PAtients With isCHEmic Heart Disease
Acronym: APACHE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Italian Society of Invasive Cardiology (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 20140003325
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Non ST Elevation Acute Coronary Syndromes; Stable Coronary Syndromes; NSTEMI; Unstable Angina
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient with non ST Elevation - Acute Coronary Syndrome
- Patient with stable Coronary Artery Disease (CAD)

SUMMARY:
An observational, retrospective, multicenter, blinded adjudication study to evaluate the clinical appropriateness of Percutaneous Coronary Intervention (PCI) indication and execution in patients with stable Coronary Artery Disease (CAD) and in patients with acute coronary syndrome without ST-segment elevation (NSTE-ACS) (ratio 4:1). Half of the included patients will be diabetic. Also the implementation of selected, key guideline recommendations will be examined.

At least 400 patients will be retrospectively selected among 22 Catheterization Laboratories in Italy in the region of Lombardia and Veneto.

This study will be conducted in compliance with Good Clinical Practices (GCP) including the Declaration of Helsinki and all applicable regulatory requirements.

DETAILED DESCRIPTION:
A strategy based on early invasive coronary angiography followed by revascularization is the most effective treatment of patients with acute coronary syndrome, especially in those with ST-segment elevation (STE-ACS). In patients with acute coronary syndrome without ST-segment elevation (NSTE-ACS), an early invasive strategy is associated with a reduction in cardiac death and myocardial infarction in patients at higher risk. In stable coronary artery disease rather no data so convincing. The undeniable evolution of techniques of PCI has been accompanied by a parallel progress of medical therapy and also from increased awareness, both cardiologists and patients, the importance of the control of coronary risk factors.

European Society of Cardiology Guide give precise indications (but often ignored) on the use of PCI or coronary artery bypass grafting according to the extent of coronary artery disease and the site of injury . However, especially in patients with NSTE-ACS often we limit ourselves to dilate the culprit stenosis, leaving untreated other injuries that underlie large myocardial territory, that is, by configuring an incomplete revascularization framework. The calculation of the SYNTAX score residual (that is, what remains after percutaneous revascularization procedure) allows to objectively verify the incompleteness of PCI treatment, which correlates with the outcome in the patient's distance . Moreover, in case of equivocal stenosis, especially in patients with stable coronary disease, large should be the use of a functional assessment using the calculation of the Fractional Flow Reserve (FFR).

This could indicate that the increase of the number of invasive diagnostic tests does not increase the number of patients with coronary artery disease extended, in which is usually indicated a surgical revascularization. So to identify patients at higher risk, may be enough specific investigations and conducted selectively.

The purpose of the pilot study APACHE is to assess the appropriateness of indication and appropriateness of execution of a sample carried out PCI in patients with stable coronary artery disease and in patients with NSTE-ACS (in the ratio 4: 1). As such, the APACHE be considered a quality improvement initiative.

Retrospective observational study, multicenter. The study population will consist of 20 cases of PCI per center (then about 400 PCI in total) selected randomly within the center of the case studies in the previous approval of the study. Of these 16 will be patients with stable coronary artery disease (including 8 with diabetes mellitus in medical therapy) and 4 will be patients with NSTE-ACS (4: 1 ratio).

Patients with a history of coronary artery bypass are excluded. The series will consist of patients in whom the procedure was carried out in the previous year to a declaration of participation in the survey and in any case after the publication of the document. There have been no previous analysis of this type in Italy and is therefore not known what is the rate of inappropriateness for PCI procedures in stable patients. It is not possible therefore to perform a calculation of sample size. However, the investigators believes that for a pilot analysis, an initial sample of 400 PCI procedures, analytically considered, is sufficient to verify the magnitude of the problem in the Italian Catheterization Laboratories.

The investigators anticipate the participation of about 20 centers in total between Lombardia and Veneto italian regions. The study will have an approximate duration of about 2 years.

The data to be collected will be different in patients with nSTE - ACS compared to patients with stable coronary artery disease. As an initiative of quality improvement, and according to extensive international literature on the subject, will not be requested individual informed consent to selected patients but only the approval of the Ethics Committee of the Center Coordinator. Patient data will be de-identified and used only in the aggregate and all individual sensitive information (name, phone, address) will be erased.

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 yrs
* Stable Coronary Artery Disease(CAD)
* Unstable Angina or NSTEMI

Exclusion criteria :

* STEMI at presentation
* previous CABG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty patients per center will be selected among those who underwent PCI in the last months, going backwards from the date of first Site visit.
  Selection will be stratified for clinical presentation in two subgroups (stable CAD:NSTEACS = 4:1) and diabetes status (1:1) for each subgroups.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with stable Coronary Artery Disease (CAD) whose clinical indication was appropriate for the treatment with Percutaneous Coronary Intervention (PCI). | 3 months
  Appropriateness will be defined by a final score of ≥ 7 of the Central Heart Team according to appropriate use criteria.

SECONDARY OUTCOMES:
Proportion of patients with complex lesions (left main, proximal LAD, three-vessel disease) treated ad hoc without documentation of Heart Team discussion in the medical records with stable CAD. | 3 months
Proportion of patients receiving incomplete revascularization (i.e. residual SYNTAX > 8)Heart Team or in patients without documented ischemia with stable CAD. | 3 months
Proportion of patients receiving guideline-recommended medical therapy at the time of PCI with stable CAD. | 3 months
Incidence of FFR-guided PCI for stenosis of uncertain significance according to the Central Heart Team or in patients without documented ischemia with stable CAD. | 3 months
Proportion of patients who received PCI but with an indication for CABG according to guidelines and no Heart team discussion in the medical record with stable CAD. | 3 months
Proportion of patients treated with PCI whose clinical indication appears appropriate defined by a final score of ≥ 7 of the Heart Team according to appropriate use criteria for Non ST elevation ACS (nSTE-ACS). | 3 months
Proportion of PCI procedures performed within 24 hours of admission in patients with nSTEACS with GRACE> 140 for nSTE-ACS. | 3 months
Proportion of patients with nSTEACS who are stabilized (no recurrent ischemic symptoms) who have multivessel disease and a high SYNTAX score (>22), without documentation of Heart Team discussion in the medical records for nSTE-ACS. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano De Servi, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo di Pavia; Sergio Leonardi, MD, Study Director — IRCCS Policlinico S. Matteo / CCRC - Cardiovascular Clinical Research Center
Locations (1):
- IRCCS Policlinico S. Matteo, Pavia, Pv, Italy

REFERENCES:
- [Result] Lucas FL, Siewers AE, Malenka DJ, Wennberg DE. Diagnostic-therapeutic cascade revisited: coronary angiography, coronary artery bypass graft surgery, and percutaneous coronary intervention in the modern era. Circulation. 2008 Dec 16;118(25):2797-802. doi: 10.1161/CIRCULATIONAHA.108.789446. Epub 2008 Dec 8. PMID 19064681
- [Result] Bauer T, Mollmann H, Weidinger F, Zeymer U, Seabra-Gomes R, Eberli F, Serruys P, Vahanian A, Silber S, Wijns W, Hochadel M, Nef HM, Hamm CW, Marco J, Gitt AK. Predictors of hospital mortality in the elderly undergoing percutaneous coronary intervention for acute coronary syndromes and stable angina. Int J Cardiol. 2011 Sep 1;151(2):164-9. doi: 10.1016/j.ijcard.2010.05.006. Epub 2010 Jun 3. PMID 20605241
- [Result] Genereux P, Palmerini T, Caixeta A, Rosner G, Green P, Dressler O, Xu K, Parise H, Mehran R, Serruys PW, Stone GW. Quantification and impact of untreated coronary artery disease after percutaneous coronary intervention: the residual SYNTAX (Synergy Between PCI with Taxus and Cardiac Surgery) score. J Am Coll Cardiol. 2012 Jun 12;59(24):2165-74. doi: 10.1016/j.jacc.2012.03.010. Epub 2012 Apr 4. PMID 22483327
- [Result] Coronary Revascularization Writing Group; Patel MR, Dehmer GJ, Hirshfeld JW, Smith PK, Spertus JA; Technical Panel; Masoudi FA, Dehmer GJ, Patel MR, Smith PK, Chambers CE, Ferguson TB Jr, Garcia MJ, Grover FL, Holmes DR Jr, Klein LW, Limacher MC, Mack MJ, Malenka DJ, Park MH, Ragosta M 3rd, Ritchie JL, Rose GA, Rosenberg AB, Russo AM, Shemin RJ, Weintraub WS; Appropriate Use Criteria Task Force; Wolk MJ, Bailey SR, Douglas PS, Hendel RC, Kramer CM, Min JK, Patel MR, Shaw L, Stainback RF, Allen JM; American College of Cardiology Foundation; American College of Cardiology Foundation Appropriate Use Criteria Task Force; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Thoracic Surgery; American Heart Association; American Society of Nuclear Cardiology; Society of Cardiovascular Computed Tomography. ACCF/SCAI/STS/AATS/AHA/ASNC/HFSA/SCCT 2012 appropriate use criteria for coronary revascularization focused update: a report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, Society for Cardiovascular Angiography and Interventions, Society of Thoracic Surgeons, American Association for Thoracic Surgery, American Heart Association, American Society of Nuclear Cardiology, and the Society of Cardiovascular Computed Tomography. J Thorac Cardiovasc Surg. 2012 Apr;143(4):780-803. doi: 10.1016/j.jtcvs.2012.01.061. PMID 22424518
- [Result] Miller FG, Emanuel EJ. Quality-improvement research and informed consent. N Engl J Med. 2008 Feb 21;358(8):765-7. doi: 10.1056/NEJMp0800136. No abstract available. PMID 18287598
- [Result] Dauerman HL. Reasonable incomplete revascularization. Circulation. 2011 May 31;123(21):2337-40. doi: 10.1161/CIRCULATIONAHA.111.033126. Epub 2011 May 16. No abstract available. PMID 21576647
- [Derived] Leonardi S, Marino M, Crimi G, Maiorana F, Rizzotti D, Lettieri C, Bettari L, Zuccari M, Sganzerla P, Tresoldi S, Adamo M, Ghiringhelli S, Sponzilli C, Pasquetto G, Pavei A, Pedon L, Bassan L, Bollati M, Camisasca P, Trabattoni D, Brancati M, Poli A, Panciroli C, Lettino M, Tarelli G, Tarantini G, De Luca L, Varbella F, Musumeci G, De Servi S. APpropriAteness of percutaneous Coronary interventions in patients with ischaemic HEart disease in Italy: the APACHE pilot study. BMJ Open. 2017 Sep 5;7(9):e016909. doi: 10.1136/bmjopen-2017-016909. PMID 28877948
- Available data/document: Report on National Journal — http://www.giornaledicardiologia.it/r.php?v=1015&a=11055&l=15130&f=allegati/01015_2012_01/fulltext/06.De%20Servi%20(47-49).pdf — De Servi S, Klugmann S: Qualità e appropriatezza dell'angioplastica coronarica in Lombardia: qualche riflessione sui dati di attivita' del registro della Società Italiana di Cardiologia Invasiva SICI-GISE) . G. Ital Cardiol 2012; 13: 47-9